CLINICAL TRIAL: NCT07309900
Title: A Single-arm, Open-label Exploratory Clinical Study of IASO208 Injection in the Treatment of Relapsed/Refractory B-cell Malignancies
Brief Title: IASO208 Injection in the Treatment of Relapsed/Refractory B-cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, MEI HENG, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IASO208CI001
Record Dates: First submitted 2025-11-26; First posted 2025-12-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory B-cell Malignancies
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IASO208 injection (Experimental)
  Interventions: Genetic: IASO208 injection

INTERVENTIONS:
Genetic: IASO208 injection — IASO208 injection is a third-generation, self-inactivated, replication-deficient Lentiviral Vector (LVV) gene therapy research drug.

SUMMARY:
This is an investigator-initiated, single-arm, open-label clinical study. It employs a dose-escalation design to evaluate the safety, pharmacokinetics, and preliminary efficacy of IASO208 injection in relapsed/refractory B-cell malignancies.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be enrolled in this study:

1. Aged ≥18 years and ≤75 years.
2. Voluntary participation in this study and signing the informed consent form.
3. Prior histopathological biopsy confirming a diagnosis of one of the following pathological types:

   * Diffuse Large B-Cell Lymphoma (DLBCL), including High-Grade B-Cell Lymphoma (HGBL);
   * Grade 3b Follicular Lymphoma (FL3b);
   * DLBCL transformed from indolent lymphoma (FL or MZL);
   * Primary Mediastinal Large B-Cell Lymphoma (PMBCL).
4. For B-cell lymphoma patients with relapsed/refractory diseases who have failed standard treatment (including relapse, non-remission, and progression), they must have received prior standard immunochemotherapy containing an anti-CD20 monoclonal antibody and an anthracycline-based regimen:

   * Relapsed disease is defined as disease relapse or progression occurring ≥12 months after the end of prior therapy.
   * Refractory disease is defined as disease progression during treatment, best response of stable disease (SD), relapse within 12 months after autologous hematopoietic stem cell transplantation, or disease progression occurring within 12 months after the end of prior therapy.
5. CD20 positivity confirmed by detection on tumor biopsy specimens obtained after the last relapse or during the screening period.
6. Presence of at least one measurable lesion according to the Lugano 2014 criteria (nodal lesion with Long Axis Diameter [LDi] >1.5 cm, extranodal lesion with LDi >1.0 cm).
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
8. Life expectancy ≥12 weeks.
9. Adequate organ function, as demonstrated by the following laboratory results

   1. Hematology: Absolute Neutrophil Count (ANC) ≥1.0 × 10⁹/L; Absolute Lymphocyte Count (ALC) ≥0.3 × 10⁹/L; Platelet count (PLT) ≥50 × 10⁹/L; Hemoglobin (Hb) ≥70 g/L (must not have received any Granulocyte Colony-Stimulating Factor [G-CSF] or Granulocyte-Macrophage Colony-Stimulating Factor [GM-CSF] treatment, or transfusion of red blood cells or platelets within 7 days prior to the laboratory assessment).
   2. Liver function: Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 3 × Upper Limit of Normal (ULN); Total Bilirubin ≤ 2 × ULN (for subjects with documented liver involvement by tumor: ALT/AST ≤5 × ULN; Total Bilirubin ≤3 × ULN).
   3. Cardiac function: Left Ventricular Ejection Fraction (LVEF) ≥50%, as measured by echocardiography or Multigated Acquisition (MUGA) scan.
   4. Oxygen saturation >92% (by pulse oximetry) at rest.
   5. Renal function: Creatinine Clearance (CrCl) ≥40 mL/min, calculated using the Cockcroft-Gault formula.
   6. Coagulation profile: Fibrinogen ≥1.0 g/L; Activated Partial Thromboplastin Time (aPTT) ≤1.5 × ULN; Prothrombin Time (PT) ≤1.5 × ULN.
10. Subjects of childbearing potential must agree to use highly effective contraceptive methods from the time of signing the informed consent form until at least 1 year after the last dose of IASO208 injection.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Subjects with central nervous system involvement.
2. Subjects who have had other malignancies within 5 years prior to screening, except for appropriately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer, ductal carcinoma in situ of the breast, or papillary thyroid carcinoma.
3. Subjects who meet any of the following conditions in infectious disease screening:

   1. Subjects positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with abnormal peripheral blood HBV DNA test (abnormal HBV DNA is defined as: quantitative detection higher than the lower limit of detection [LLD], above the normal range, or positive qualitative detection).
   2. Subjects positive for hepatitis C virus (HCV) antibody with positive peripheral blood HCV RNA.
   3. Subjects positive for human immunodeficiency virus (HIV) antibody.
   4. Subjects with syphilis.
   5. Subjects with active cytomegalovirus (CMV) infection.
4. Uncontrolled active bacterial, fungal, or viral infection prior to enrollment, as evidenced by:

   1. Persistent infection-related symptoms/signs requiring intravenous anti-infective therapy; or
   2. No improvement in clinical symptoms or examinations after appropriate anti-infective therapy.
5. Severe cardiac diseases, including but not limited to: unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] Class ≥ III), or severe arrhythmia.
6. History of central nervous system diseases or disorders within 6 months prior to screening, such as epilepsy, paralysis, aphasia, cerebral infarction, cerebral hemorrhage, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome (e.g., cerebral aneurysm, epilepsy, stroke [except for lacunar infarction], dementia, psychosis), or subjects with impaired consciousness.
7. Previous solid organ transplantation.
8. Previous allogeneic hematopoietic stem cell transplantation (allo-HSCT), allogeneic CAR-T therapy, or other allogeneic donor adoptive cell therapies.
9. Subjects who do not meet the required washout periods for the following prior therapies/treatments before enrollment:

   1. Cytotoxic chemotherapy, monoclonal antibodies, bispecific antibodies, or antibody-drug conjugates (ADCs) within 4 weeks prior to enrollment.
   2. Ongoing requirement for systemic corticosteroids or other immunosuppressive therapy within 4 weeks prior to enrollment.
   3. Radiotherapy or major surgery of Grade 4 severity within 4 weeks prior to enrollment; or planned general anesthesia surgery within 12 weeks after receiving the study treatment.
   4. Vaccination or treatment with any investigational products within 4 weeks prior to enrollment.
   5. Autologous hematopoietic stem cell transplantation or autologous CAR-T therapy within 12 weeks prior to enrollment.
10. Presence of other unstable systemic diseases, as determined by the investigator, including but not limited to severe hepatic, renal, or metabolic diseases requiring treatment.
11. Adverse events from previous anti-tumor therapies have not resolved to baseline or Grade ≤ 2 (excluding alopecia, fatigue, and peripheral neuropathy).
12. Known history of hypersensitivity to any excipient component of the IASO208 injection.
13. Pregnant or lactating women.
14. Any other condition deemed by the investigator as inappropriate for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2028-12-15 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicity (DLT); | Up to 28 days from dosing
  Percentage of participants who experienced DLT within 28 days after IASO208 administration.
The incidence and severity of adverse events (AEs) | Up to 2 years from dosing
  Percentage of participants who experienced AEs after IASO208 administration and severity was graded according to the NCI-CTCAE version 5.0.
The types、incidence and severity of abnormal laboratory tests; | Up to 2 years from dosing
  The types、incidence and severity of abnormal laboratory results assessed by CTCAEV5.0 will be analyzed and reported.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years from dosing
  ORR was defined as the percentage of participants who achieved partial response (PR) or better as assessed by the investigator according to the Lugano 2014 Criteria.
Objective response rate (ORR) at pre-specified timepoints | Up to 2 years from dosing
  ORR at 3, 6, 12 months as assessed by the investigator according to the Lugano 2014 Criteria.
Complete response rate (CRR) | Up to 2 years from dosing
  CRR was defined as the percentage of participants who achieved complete response (CR) as assessed by the investigator according to the Lugano 2014 Criteria.
Duration of Response (DOR) | Up to 2 years from dosing
  DOR was defined as the time (in months) from the date of initial documented response (PR or better response) to the date of first documented evidence of progressive disease (PD) or death.
Time to Response (TTR) | Up to 2 years from dosing
  TTR was defined as the time between date of IASO208 administration and the first efficacy evaluation that the participant met all criteria for PR or better.
Progression-free Survival (PFS) | Up to 2 years from dosing
  PFS was defined as the time from the date of IASO208 administration to the date of first documented disease progression or death.
Overall Survival (OS) | Up to 2 years from dosing
  OS was defined as the time from the date of IASO208 administration to the date of the participant's death.
Maximum concentration (Cmax) of viral particle titer in peripheral blood following IASO208 administration | Up to 7 days from dosing
  Cmax of viral particle titer in peripheral blood will be observed and calculated.
Peak time (Tmax) of viral particle titer in peripheral blood following IASO208 administration | Up to 7 days from dosing
  Tmax of viral particle titer in peripheral blood will be observed and analyzed.
Area under the concentration-time curve from day 0 to day 7 (AUC0-7) of viral particle titer in peripheral blood following IASO208 administration | Up to 7 days from dosing
  AUC0-7d refers to the area under the concentration-time curve from day 0 (IASO208 dosing moment) to day 7 .
Concentration of vector copy numbers (VCN) in peripheral blood | Up to 2 years from dosing
  Concentration of VCN will be measured and reported following IASO208 administration.
CAR-T cell count in peripheral blood | Up to 2 years from dosing
  Concentration of CAR-T cell count will be observed and reported following IASO208 administration.
B lymphocytes in peripheral blood | Up to 2 years from dosing
  Concentration of B lymphocytes in peripheral blood will be observed following IASO208 administration.
Cytokines in peripheral blood | Up to 2 years from dosing
  Cytokines not limited to CRP、Ferritin 、、IL-6、IFN-γ、TNF-α in peripheral blood will be observed following IASO208 administration.

OTHER OUTCOMES:
Percentage of participants with positive anti-drug antibodies (ADA) | Up to 2 years from dosing
  Percentage of participants with positive antibodies will be reported.
Percentage of participants with Replication-Competent Lentivirus (RCL) | Up to 15 years from dosing
  Percentage of participants with RCL will be reported.
Percentage of participants with detectable viral particles in secretions following IASO208 administration. | Up to 2 years from dosing
  Percentage of participants with detectable viral particles in secretions will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No